CLINICAL TRIAL: NCT05108506
Title: To Void or Not to Void After Same-day Discharge, Non-urogynecologic, Minimally Invasive Hysterectomy, That is the Question
Brief Title: Strict Need to Void After Same-day Discharge, Non-urogynecologic, Minimally Invasive Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00307084
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Urinary Retention Postoperative
Keywords: Minimally invasive hysterectomy; Urinary retention; Some day discharge
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No strict need to void following surgery before discharge (Experimental): Participants randomized to this arm will have no strict need to void following surgery before they are discharged.
  Interventions: Behavioral: No Strict need to void following surgery
- Strict need to void following surgery before discharge (Placebo Comparator): Participants randomized to this arm will have a strict need to void following surgery before they are discharged.
  Interventions: Behavioral: Strict need to void following surgery

INTERVENTIONS:
Behavioral: No Strict need to void following surgery — Certain patient will be randomized without a strict need to void prior to discharge following surgery.
  Arms: No strict need to void following surgery before discharge
Behavioral: Strict need to void following surgery — Certain patient will be randomized with a strict need to void prior to discharge following surgery.
  Arms: Strict need to void following surgery before discharge

SUMMARY:
Patients who are undergoing non-urogynecologic, minimally invasive (laparoscopic, robotic) hysterectomy who are discharged the day of surgery will be randomized to a strict need to void versus no need to void prior to discharge.

To determine if a strict versus liberal voiding trial following the aforementioned surgery in same day discharge patients increases rates of post-operative urinary retention, urinary tract infection (UTI), or re-presentation and if there is a difference in Post-Anesthesia Care Unit (PACU) time and costs.

ELIGIBILITY:
Inclusion Criteria:

* Women 18+ undergoing minimally invasive benign, non-urogynecologic hysterectomy
* English speaking

Exclusion Criteria:

* At the surgeons discretion based on amount of bladder dissection the patient can be removed from the study at the conclusion of surgery
* Any patient with a history of prior urologic procedures
* Patients with any baseline known urinary disease
* Any bladder injury at the time of surgery
* Any combined cases with other surgical services
* Patients undergoing surgery for prolapse or incontinence symptoms
* Patients who are ultimately not discharged the same day and remain in house overnight

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Amount of time spent in PACU | 2 years
  This will assess the amount of time spent (in hours) in PACU.

SECONDARY OUTCOMES:
Rates of urinary retention | 2 years
  Will measure rates of urinary retention.
Rates of UTI | 2 years
  Will measure rates of UTI.
Rates of re-presentation to the ER | 2 years
  Will measure rates of re-presentation to ER.
Cost of stay in PACU | 2 years
  This will assess the cost pertaining to the time spent in the PACU to determine if the time spent has a significant impact on the cost.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Patzkowsky, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No